CLINICAL TRIAL: NCT04226313
Title: Cervical Cancer Prevention Using Self-sampling and Human Papillomavirus Detection
Brief Title: Self-sampling for Non-attenders to Cervical Cancer Screening
Acronym: KOPRETINA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Institute of Molecular and Translational Medicine, Czech Republic (Other)
Collaborators: National Institute for Cancer Research, Czech Republic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 5850
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Cervical Cancer; Cervical Dysplasia; Human Papillomavirus Infection
Keywords: human papillomavirus; HPV; self-sampling; cervicovaginal swab; cervical cancer screening; non-attendance
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia; Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Self-sampling device sent at home (Active Comparator): Women randomly selected from a commercial vendor database (both attenders and non-attenders) receive a mail inviting them to perform a cervicovaginal self-sampling at their home (with the device provided). Returned self-sampled swabs will be tested by CE-IVD-marked (Conformité Européenne, In Vitro Diagnostics) HPV diagnostic test validated for use in primary cervical cancer screening. The arm will include approx. 5000 participants.
  Interventions: Diagnostic Test: Self-sampling by Evalyn Brush
- Self-sampling device sent by gynecologist(s) (Experimental): Women selected from databases of cooperating gynecologists (non-attenders for at least 3 years) receive a mail inviting them to perform a cervicovaginal self-sampling at their home (with the device provided). Returned self-sampled swabs will be tested by CE-IVD-marked HPV diagnostic test validated for use in primary cervical cancer screening. The arm will include approx. 5000 participants.
  Interventions: Diagnostic Test: Self-sampling by Evalyn Brush
- Self-sampling device obtained from general practitioner(s) (Experimental): Women selected from databases of cooperating general practitioners (non-attenders for at least 3 years) receive a self-sampling device. Returned self-sampled swabs will be tested by CE-IVD-marked HPV diagnostic test validated for use in primary cervical cancer screening. The arm will include approx. 5000 participants.
  Interventions: Diagnostic Test: Self sampling by Evalyn Brush home or in GP´s clinic

INTERVENTIONS:
Diagnostic Test: Self-sampling by Evalyn Brush — Women will perform a cervicovaginal self-sampling at their home using Evalyn Brush.
  Arms: Self-sampling device sent at home; Self-sampling device sent by gynecologist(s)
Diagnostic Test: Self sampling by Evalyn Brush home or in GP´s clinic — Women will perform a cervicovaginal self-sampling at their home or the GP´s clinic using Evalyn Brush
  Arms: Self-sampling device obtained from general practitioner(s)

SUMMARY:
The trial will evaluate whether self-sampling and human papillomavirus (HPV) testing may increase cervical cancer screening attendance among under-screened women in Czech Republic. Different ways of offering self-sampling device will be evaluated.

DETAILED DESCRIPTION:
Despite the existence of an effective cervical cancer screening in the Czech Republic, cervical cancer is the cause of about 800 new cases and 400 deaths every year. One of the major problem of the Czech cervical cancer screening is low participation. An effective strategy to increase cervical cancer screening attendance is one of the main challenges. The offering of self-sampling to the cervical cancer screening non-attenders could increase women's participation as was shown in several European countries.

The trial should determine acceptability of the self-sampling followed by HPV DNA test by Czech women and therefore usability of the self-sampling device to increase cervical cancer screening attendance among under-screened women. Three different approaches will be tested: women will receive a self-sampling device by mail (Arm A); receive a self-sampling device by gynecologist (Arm B); receive a self-sampling device by general practitioner (Arm C). Comparisons of the screening attendance among the arms will be made. To address also potential effects on inequities, the analyses will include comparisons by sociodemographic characteristics. Women from the database of commercial vendor will be included to the Arm A regardless of whether or not they participate in cervical cancer screening program. Women who do not participate in cytology-based cervical cancer screening program for at least three years will be included through their gynecologist (Arm B) or general practitioner (Arm C) database.

The second focus of the trial is the evaluation of high-risk human papillomavirus prevalence in screening population of Czech women (attenders and non-attenders of cervical cancer screening) since there are no relevant data for the Czech Republic. Study participants may volunteer for archiving of remaining biological materials for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Women with age 30-65 years; for arm A women > 65 years are allowed
* Women live in the Czech Republic.
* Women who have not participate in cervical cancer screening program in the Czech Republic for at least 3 years (Arm B and C).
* Women with completed informed consent.
* Women capable of self-sampling of cervicovaginal swab.

Exclusion Criteria:

* Pregnant women.
* Women with no sexual intercourse experience.
* Women after hysterectomy including cervix.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 15000 (Estimated)
Dates: Start 2019-09-23 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Screening participation | 12 months
  Comparison of the percentages of women who return a cervicovaginal swab sampled by self-sampling device in different arms of the study. Identification of the best approach to address women who do not participate in standard cervical cancer screening program
Prevalence of high-risk HPV | 12 months
  Evaluation of the prevalence of high-risk human papillomavirus infection in screening population of Czech women within different arms of the study (attenders/non-attenders).

SECONDARY OUTCOMES:
Sociodemographic characteristics | 12 months
  Comparison the distribution of sociodemographic characteristics (education, age, place of residence) and reasons for previous non-attendance for screening by intervention and attendance status in women who return a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Marian Hajduch, MD, PhD., Study Director — IMTM, Palacky University in Olomouc, Faculty of Medicine and Dentistry
Locations (1):
- University Hospital Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: No